CLINICAL TRIAL: NCT04904978
Title: Evaluation of Two Different Toothpastes for the Clinical Management of Extrinsic Stains: Randomized Clinical Trial.
Brief Title: Evaluation of Two Different Toothpastes for Clinical Management of Extrinsic Stains.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-BLANKSBLACK
Record Dates: First submitted 2021-05-22; First posted 2021-05-27 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Extrinsic Staining of Tooth - Medication
Keywords: toothpaste; extrinsic stains

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Use of Blanx Black Toothpaste
  Interventions: Other: Blanx Black Toothpaste
- Control Group (Active Comparator): Use of Colgate Sensation White toothpaste.
  Interventions: Other: Colgate Sensation White

INTERVENTIONS:
Other: Blanx Black Toothpaste — Use of Blanx Black Toothpaste twice a day per at least 2 minutes.
  Arms: Trial Group
Other: Colgate Sensation White — Use of Colgate Sensation White Toothpaste twice a day per at least 2 minutes
  Arms: Control Group

SUMMARY:
The aim of the study is to assess the efficacy of Blanx Black Toothpaste against extrinsic stains of teeth.

Patients who sign the informed consent will participate to the study.

At the baseline, the collection of Plaque Index, modified Lobene index and Bleeding Index will be performed, giving the instruction for a proper home oral hygiene. Professional supragingival and subgingival dental hygiene with piezoelectric will be performed. Then, patients will be randomly divided into two groups:

* Trial Group will use Blanx Black Toothpaste (2 minutes brushing) twice a day for the all the study duration;
* Control Group will use Colgate Sensation White Toothpaste (2 minutes brushing) twice a day.

Patients will be reevaluated after 10 days, after 1 month and after 3 months, collecting again the indices and improving home oral care.

DETAILED DESCRIPTION:
The aim of the study is to assess the efficacy of Blanx Black Toothpaste against extrinsic stains of teeth.

For this purpose, patients addressing to the Dental Hygiene Unit that agree to participate to the study will be enrolled after signing the informed consent.

At the baseline, the collection of Plaque Index, modified Lobene index and Bleeding Index will be performed, giving the instruction for a proper home oral hygiene. Professional supragingival and subgingival dental hygiene with piezoelectric will be performed. Then, patients will be randomly divided into two groups:

* Trial Group will use Blanx Black Toothpaste (2 minutes brushing) twice a day for the all the study duration;
* Control Group will use Colgate Sensation White Toothpaste (2 minutes brushing) twice a day.

Patients will be reevaluated after 10 days, after 1 month and after 3 months. After the reinforcement of home oral hygiene, the above mentioned indices will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presence of extrinsic stains
* Patients with high compliance

Exclusion Criteria:

* Underage patients
* Patients suffering from neurological or psychiatric disorders
* Pregnant women
* Patients undergoing anticancer chemotherapy
* Patients with low compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Change in BOP - Bleeding on Probing (percentage) | Baseline, 10 days, 1 month, 3 months
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  Percentage of sites with bleeding on probing determines the BOP%.
Change in MLI - Modified Lobene Index | Baseline, 10 days, 1 month, 3 months
  The facial surface of each anterior tooth was divided into two regions. The first is the gingival region which was a crescent-shaped band of the labial surface about 2 mm wide adjacent to the free margin of the gingiva and extending to the crest of the interdental papillae of the adjacent teeth. The second is the body region which constitutes the remainder of the labial surface of the tooth.
  The gingival and body regions were scored separately.
  Intensity - Scoring criteria:
  * 0: no stain;
  * 1: mild stain, from yellow to light brown or gray;
  * 2: mild stain, brown colored;
  * 3: heavy stain, from dark brown to black.
  Area - Scoring criteria:
  * 0: no stain;
  * 1: 1/3 extension of the stain;
  * 2: from 1/3 to 2/3 extension of the stain;
  * 3: stain covering over two-thirds of the region. stain extent.
Change in Plaque Control Record (PCR%) | Baseline, 10 days, 1 month, 3 months
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.Scoring criteria:
  * 0: no bleeding
  * 1: mild bleeding
  * 2: severe bleeding The number of bleeding sites is divided per the total number of probed sites; the ratio is multiplied X 100.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.